CLINICAL TRIAL: NCT05748496
Title: A Pilot Study to Evaluate Efficacy of Brief Behavioral and Sleep Hygiene Education With Mindfulness Intervention on Sleep Duration, Sleep Timing, Sleep Quality, Anxiety, Depression, and Quality of Life in Adolescents
Brief Title: Study to Evaluate Efficacy of Brief Behavioral and Sleep Hygiene Education With Mindfulness Intervention on Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solveig Magnusdottir (Other Government)
Collaborators: MyCardioLLC (Unknown)
Responsible Party: Sponsor-Investigator, Solveig Magnusdottir, Medical Doctor, Akureyri Hospital
Organization: Akureyri Hospital (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VSN-22-174
Record Dates: First submitted 2023-02-20; First posted 2023-02-28 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Brief behavioral sleep therapy, sleep hygiene education and mindfulness training
- Controle (No Intervention)

INTERVENTIONS:
Behavioral: Brief behavioral sleep therapy, sleep hygiene education and mindfulness training — Brief behavioral sleep therapy, sleep hygiene education and mindfulness training using breathing exercises and Yoga Nidra
  Arms: Intervention

SUMMARY:
Sleep plays a fundamental role in both mental- and physical-health, with good sleep health including adequate duration and quality, appropriate timing, regularity, and absence of sleep disorders. The purpose of this study is to evaluate sleep in adolescent and if brief behavioral and sleep hygiene education with mindfulness intervention improves, sleep timing, sleep duration, sleep quality, anxiety/depression, and quality of life.

During adolescence extensive physiological changes happen that make it easier for adolescents to stay up later, that may increase the time it may take them to fall-asleep and developing insomnia symptoms. At the same time psychosocial changes happen, that may may even have been further amplified in the last decade, with increase in social media use and evening screen-time. As sleep need is not decreased and with adolescents having to wake up at "socially acceptable times" rather than the endogenous sleep offset time, sleep duration may be shortened causing chronic sleep loss and daytime sleepiness. Insufficient sleep in adolescents may affect their daytime functioning, causing fatigue and memory issues, affect school attendance and academic performance, affect mood, mental- and physical health, cause behavioral dysfunction and has been associated with worse health outcomes, adverse risk behaviors and even increase risk for accidents.This study should advance understanding of sleep in adolescents and if this simple interventions can be effective in improving their sleep and mental health. If effective larger studies will be needed to evaluate if there might be a value in implementing changes in the infrastructure of the educational system to better support sleep and mental health of adolescent.

DETAILED DESCRIPTION:
The study is a prospective cross-sectional study implementing a brief behavioral and sleep hygiene education with mindfulness intervention in adolescents in the age-range of 16-19-years interested to participate and willing to sign a consent. Sleep duration, sleep timing and sleep quality will be measured with objective home sleep test for three (3) week-nights and two (2) weekend-nights and sleep, anxiety and depression symptoms will be evaluated with subjective questionnaires before starting the 4-week intervention. After the 4-week intervention sleep, anxiety and depression symptoms will be evaluated again using both the objective home sleep test and questionnaires to measure if the intervention improved sleep timing, duration and/or quality as well as symptoms of anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

Students interested to participate and able to sign enlightened consent

Exclusion Criteria:

Atrial fibrillation or ventricular trigeminy Severe and uncontrolled asthma or severe pulmonary disease Moderate and severe obstructive sleep apnoea (OSA)

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
To evaluate if changes will be observed in sleep quality measured with sleep quality index (SQI) | 4-week intervention
  Intervention with brief behavioral and sleep hygiene education and mindfulness training with breathing exercises and Yoga Nidra
To evaluate if changes will be observed in sleep timing and duration (hours, minutes) | 4-week intervention
  Intervention with brief behavioral and sleep hygiene education and mindfulness training with breathing exercises and Yoga Nidra

SECONDARY OUTCOMES:
To evaluate if changes will be observed in anxiety evaluated using the General Anxiety Disorder-7 scale (score 0-21) | 4-week intervention
  Intervention with brief behavioral and sleep hygiene education and mindfulness training with breathing exercises and Yoga Nidra

CONTACTS AND LOCATIONS:
Overall Officials: Solveig Magnusdottir, MD, Principal Investigator — MyCardioLLC
Locations (1):
- Menntaskolinn a Akureyri, Akureyri, Iceland

IPD SHARING:
Plan to Share IPD: No